CLINICAL TRIAL: NCT02898506
Title: Incretin-based Therapy in Late Preclinical Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Riitta Veijola, Professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LiraAABDG10-30; 2014-004761-25 (EudraCT Number); U1111-1177-0704 (Other: WHO); 3-SRA-2014-301-M-R (Other Grant/Funding Number: Juvenile Diabetes Research Foundation International)
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Type 1; Diabetes, Insulin-Dependent; Liraglutide; Preclinical Type 1 Diabetes; GLP-1 Analogue; Dysglycemia; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): Subjects with multiple islet autoantibodies and dysglycemia and aged 10-30 years are treated with Victoza®
  Interventions: Drug: Victoza®
- Placebo (Placebo Comparator): Subjects with multiple islet autoantibodies and dysglycemia and aged 10-30 years are treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Victoza® — Daily subcutaneous injections with increasing doses up to 1.8 mg per day. Duration of treatment 6 months and thereafter follow-up of 6 months.
  Arms: Liraglutide
Drug: Placebo — Daily subcutaneous injections with increasing doses up to 1.8 mg per day. Duration of treatment 6 months and thereafter follow-up of 6 months.
  Arms: Placebo

SUMMARY:
The objective of the trial is to study whether daily treatment with liraglutide improves endogenous insulin secretion, postpones progression to overt Type 1 diabetes, and is tolerable and safe in subjects aged 10-30 years, who are positive for multiple islet autoantibodies and have dysglycemia.

ELIGIBILITY:
Inclusion Criteria:

* 10-30 years of age
* positive for at least 2 islet autoantibodies
* glucose intolerance or dysglycemia: impaired glucose tolerance (IGT, 2-hour p-gluc 7.8-11.0mmol/l), or impaired fasting glucose (IFG, fp-gluc 6.1-6.9mmol/l), and/or 10% rise in HbA1c since the last measurement (2 - 12 mo ago), and/or p-gluc at least 11.1mmol/l at 30, 60 or 90 min during OGTT
* not pregnant

Exclusion Criteria:

* allergic to liraglutide or other ingredients of Victoza
* type 1 diabetes
* diabetic ketoacidosis
* previous treatment in the last three months with any antidiabetic medication
* impaired liver or kidney function or on dialysis
* severe heart failure
* severe stomach or gut problem resulting in gastroparesis, or inflammatory bowel disease
* past or current history of pancreatitis
* serum calcitonin value above normal (>50 ng/l or at least 3.4pmol/l)
* presence of any chronic metabolic, hematologic or malignant disease
* obesity BMI at least 30
* pregnant females and females of childbearing potential who are not using adequate contraceptive methods.
* breast-feeding

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
FPIR (1+3min serum insulin level after iv glucose infusion) | 12 months
  First phase insulin response during 10-min IVGTT (intravenous glucose tolerance test)

SECONDARY OUTCOMES:
Safety: serum and urine amylase, serum lipase, serum calcitonin, hypoglycemia | 12 months
  Safety: serum and urine amylase, serum lipase, serum calcitonin, hypoglycemia
Tolerability | 12 months
  Tolerability: frequency of side effects, hypoglycaemia and gastrointestinal symptoms in particular
Serum C-peptide AUC | 12 months
  Serum C-peptide area under the curve (AUC) during 2-hour OGTT (oral glucose tolerance test)

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Veijola, MD, Principal Investigator — University of Oulu
Locations (4):
- Finland (3):
  - University of Oulu and Oulu University Hospital, Dept of Children and Adolescents, Oulu
  - University of Tampere and Tampere University Hospital, Tampere
  - University of Turku and Turku University Hospital, Turku
- Lund University and Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Kero J, Koskenniemi JJ, Karsikas S, Pokka T, Lou O, Toppari J, Veijola R. INnoVative trial design for testing the Efficacy, Safety and Tolerability of 6-month treatment with incretin-based therapy to prevent type 1 DIAbetes in autoantibody positive participants: A protocol for three parallel double-blind, randomised controlled trials (INVESTDIA). Diabet Med. 2022 Oct;39(10):e14913. doi: 10.1111/dme.14913. Epub 2022 Jul 22. PMID 35797241